CLINICAL TRIAL: NCT00314769
Title: Long-Term Improvement in Training Effects by Transcranial DC Stimulation
Brief Title: Long-Term Improvement in Motor Learning by Transcranial Direct Current Stimulation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060138; 06-N-0138
Record Dates: First submitted 2006-04-13; First posted 2006-04-14 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-12-16

CONDITIONS: Healthy Volunteers
Keywords: Transcranial Direct Current Stimulation (TDCS); Motor Learning; Transcranial Magnetic Stimulation (TMS); Cortical Re-Organization; Neuroplasticity; Neurorehabilitation; TBI; Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
This study will examine whether continuous use of transcranial direct current stimulation (tDCS) in combination with motor training can lead to long-term improvement in movement performance beyond what can be achieved with motor training alone.

Healthy normal volunteers 18-80 years of age who are clearly right- or left-handed may be eligible for this study. Each candidate is screened with a medical history, clinical and neurological examination, questionnaires to evaluate memory, attention, and handedness and a brain MRI, if one has not been done by NINDS within 12 months of entering the study. Pregnant women may not participate.

The study involves 10 sessions (in addition to the screening visit) over 3 months. Sessions 1-5 are completed over 5 consecutive days. Sessions 6-10 are divided over the remaining time. Participants are randomly assigned to one of three groups: 1) tDCS during motor training; 2) tDCS after training; or 3) training with sham tDCS. During these sessions, participants perform a pinch force task (squeezing a small device between the thumb and forefinger) and visuomotor tasks (using a device to move the cursor on a computer screen to various targets and holding the cursor in place for 1 second).

During the motor training and performance sessions, participants have the following procedures.

* TMS measurements: A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil.
* tDCS: Small, wet sponge electrodes are applied to the head - one above the eye and the other on the back of the head. A small electrical current is passed between them. The subject may feel an itching or tingling sensation under the electrodes or see light flashes. Some sessions are done with sham tDCS.
* Surface electromyography: Electrodes are filled with a conductive gel and taped to the skin over one small hand muscle to measure the electrical activity of muscles.
* Behavioral measurements: Evaluation of learned movement tasks
* Questionnaires to evaluate the subject's attention, fatigue and mood before and after testing

DETAILED DESCRIPTION:
OBJECTIVES:

Motor practice and use over one session leads to use-dependent plasticity. When practice is repeated over multiple sessions, motor performance continues improving until a plateau in performance, the so-called ceiling effect is reached. This issue is particularly important in neurorehabilitative treatments in which patients usually reach a ceiling effect without further improvement. Thus, it would be desirable to modify ceiling effects in motor rehabilitation. The purpose of this protocol is to determine if repeated applications of TDCS, a form of non-invasive cortical stimulation known to transiently improve performance, in association with training, could elicit additional improvements in motor performance beyond the ceiling effect identified during performance of a visuomotor training task.

We will test the hypothesis that anodal TDCS applied over M1 in temporal relation with motor training will lead to more prominent long-term learning of a visuomotor task relative to sham stimulation (which would document the ceiling effect) in healthy individuals and chronic stroke patients and traumatic brain injury (TB1) patients..

STUDY POPULATION:

We plan to study 177 healthy volunteers (part 1) and 60 chronic stroke patients (part 2) and 50 TB1 patients with 50 additional healthy volunteers (part 3). Therefore, an overall enrollment of 337 participants is planned.

DESIGN:

The study will follow a parallel design. Healthy volunteers (part 1) and stroke patients (part 2)will be randomly allocated to one of three groups. Each group will receive anodal TDCS or sham in a fixed time frame related to motor training (during or immediately after motor training). TB1 patients and healthy volunteers (part 3) will be randomly allocated to one of two groups. Each group will receive either sham or anodal tDCS during training.

Healthy volunteers and stroke patients will participate in 10 sessions. First, they will train a visuomotor task (VMT) on 5 consecutive days while receiving sham stimulation (group 3) or TDCS during (group 1), or immediately after (group 2) the training. Performance of the VMT will be re-evaluated at 30, 60 and 90 days after the first training session.

Traumatic brain injury (TB1) patients and a group of healthy volunteers (part 3) will participate in 6 sessions. First, they will train a visumomotor task (VMT) on 3 consecutive days while receiving anodal tDCS or sham stimulation during the training. Performance of the VMT will be re-evaluated at 30, 60, and 90 days after the first training session.

OUTCOME MEASURES:

Primary outcome measure will be the percentage change (from baseline to day 8 in healthy volunteers and stroke patients, and from baseline to day 3 in traumatic brain injury) in the total time necessary to complete 15 correct trials of the visuomotor task.

Secondary outcome will be accuracy (no. of errors) and timing (speed) variability of force adaptation in the visuomotor task (Celnik, own data), and pinch force at all other time points, including day 5 as a measure of learning over the training period and 3 months as a measure for long-term retention. In the patient group the Jebsen Taylor Test will be used to assess gross motor function. To better understand the mechanisms underlying the proposed behavioral gains, we will use single- and paired pulse transcranial magnetic stimulation (TMS) to identify corticomotor excitability changes. Furthermore the volunteers will answer several questionnaires to evaluate fatigue and mood (PANAS) and perform short neuropsychological control task to control for changes in attention and memory function.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include HEALTHY VOLUNTEERS under the following circumstances:

1. Age of 18 to 80 years.
2. Written informed consent is given by the participant.
3. Mini-Mental-Status examination greater than 23 points.
4. Handedness as assessed by Edinburgh handedness inventory shows a laterality index (LI) greater than 75 (dexterity) or LI of less than -75 (left-handedness).
5. Ability to concentrate and to perform the tasks required in the present study.
6. Commitment to participate in the long-term follow-up (up to 3 months).

We will include STROKE PATIENTS under the following circumstances:

1. Age of 18 to 80 years.
2. Stroke more than 3 months ago.
3. Single stroke with hemispheric lesions.
4. Stroke that affected one side of the brain (unilateral stroke).
5. Patients with initially severe motor paresis (below MRC grade 2), who subsequently recovered to the point that they have a residual motor deficit but still able to perform the tasks required by the study.
6. Commitment to participate in the long-term follow-up (up to 3 months).
7. Written informed consent is given by the patient.
8. Mini-Mental-Status examination greater than 23 points.
9. Handedness as assessed by Edinburgh handedness inventory shows a laterality index (LI) greater than 75 (dexterity) or LI of less than -75 (left-handedness).

We will include TBI PATIENTS under the following circumstances:

1. Age of 18 to 80 years
2. Handedness as assessed by Edinburgh handedness inventory showing a laterality index (L1) greater than 75 (dexterity) or L1 of less than -75 (left-handedness)
3. Ability to concentrate on a computer task for up to an hour.
4. Ability to perform dominant hand thumb opposition against resistance.
5. Willingness to commit to the time involved in the study.
6. Willingness and ability to give consent.
7. TBI occurred from non-penetrating blunt, acceleration, or deceleration forces to the head.
8. TBI is of mild to moderate severity, based on loss of consciousness up to 24 hours, post-traumatic amnesia up to 7 days, or GCS score (9-15), as can be ascertained by medical records or patient report.
9. TBI more than 6 months ago

EXCLUSION CRITERIA:

We will exclude healthy volunteers and stroke patients, and TBI patients if one of the following conditions applies:

1. Unable to perform the tasks.
2. A history of severe neurological illness, e.g. brain tumor, epilepsy or a history of symptomatic seizures, polyneuropathy etc.
3. A history of severe alcohol or drug abuse, psychiatric illness such as severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).
4. More than moderate uncontrolled medical problems (e.g. active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, hypo/hyperthyroidism, severe diabetes, peripheral arteriopathy, or a deteriorated condition due to age, or other medical conditions as determined by the study physician, that would interfere with participation in this study).
5. Increased intracranial pressure as evaluated by clinical means (presence of papilledema in eye ground exam, compressed sulci/ventricle on MRI scan).
6. Metal in the body which might make having an MRI unsafe (e.g., vascular clips, cochlear implant) in the cranium (except in the mouth), pacemaker, implanted medication pumps, neural stimulators.
7. Drug treatment acting primarily on the central nervous system which lowers the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants (for the TMS component only).
8. Any visual disturbances, especially visual acuity less than 60%.
9. Diseased or damaged skin over the face or scalp.
10. Acute or chronic tendosynovitis, severe rheumatoid arthritis, active joint deformity of arthritic origin, according to the hand.
11. Professionally practiced playing a musical instrument or trained as a typist.
12. Pregnancy (for the MRI component only).

    EXCLUSION CRITERIA - FOR STROKE PATIENTS ONLY:
13. Both sides of the brain are affected by the stroke or clear bilateral motor impairment.

    EXCLUSION CRITERIA - FOR TBI PATIENTS ONLY:
14. TBI from penetrating gunshot or explosive trauma.
15. Post-traumatic seizures
16. No reported changes in both the Glascow Coma Scale and mental status following injury.
17. Active depression of any severity with psychoactive medication changes in the last 2 months.
18. Active psychosis, disruptive or violent behavior, or poor motivational capacity.
19. Pending litigation regarding the trauma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-04-07; Study Completion 2013-12-16

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Butefisch CM, Davis BC, Wise SP, Sawaki L, Kopylev L, Classen J, Cohen LG. Mechanisms of use-dependent plasticity in the human motor cortex. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3661-5. doi: 10.1073/pnas.97.7.3661. PMID 10716702
- [Background] Karni A, Meyer G, Rey-Hipolito C, Jezzard P, Adams MM, Turner R, Ungerleider LG. The acquisition of skilled motor performance: fast and slow experience-driven changes in primary motor cortex. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):861-8. doi: 10.1073/pnas.95.3.861. PMID 9448252
- [Background] van Mier H, Tempel LW, Perlmutter JS, Raichle ME, Petersen SE. Changes in brain activity during motor learning measured with PET: effects of hand of performance and practice. J Neurophysiol. 1998 Oct;80(4):2177-99. doi: 10.1152/jn.1998.80.4.2177. PMID 9772270